CLINICAL TRIAL: NCT03833466
Title: Metformin in Combined With Cisplatin Plus Paclitaxel as Neoadjuvant Therapy With Advanced Esophageal Squamous Cell Carcinoma (ESCC)
Brief Title: Metformin in Combined With Cisplatin Plus Paclitaxel With Advanced Esophageal Squamous Cell Carcinoma (ECMTPneo)
Acronym: ECMTPneo
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shen Lin, Clinical Professor, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESCC-MTPneo
Record Dates: First submitted 2019-01-22; First posted 2019-02-07 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Advanced Esophageal Squamous Cell Carcinoma; Neoadjuvant Therapy; Metformin; Cisplatin; Paclitaxel
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Metformin; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- metformin and chemotherapy (Experimental)
  Interventions: Drug: metformin and chemotherapy

INTERVENTIONS:
Drug: metformin and chemotherapy — Drug: Metformin Metformin is orally administered as 500mg bid for 7 days and escaladed to 500mg tid if adverse events are tolerated.
  Drug: Cisplatin Cisplatin is given at 75mg/m2 intravenously on day 1 of each 21 day cycle.
  Drug: Paclitaxel Paclitaxel is given at 175mg/m2 intravenously on day 1 of each 21 day cycle.

SUMMARY:
This is an open-label phase II trial investigating the effect of metformin in combined with cisplatin plus paclitaxel as neoadjuvant therapy with advanced esophageal squamous cell carcinoma.

DETAILED DESCRIPTION:
In this prospective phase II study, eligible patients are received cisplatin plus paclitaxel for 2-4 cycles combined with metformin orally. The investigators aim to compare the tumor metabolic pathway and tumor microenvironment of pre-chemotherapy endoscopic biopsy samples and post-chemotherapy surgical resection samples.

ELIGIBILITY:
Inclusion Criteria:

* Having signed informed consent.
* Age 18 to 70 years old
* Histologically confirmed esophageal squamous carcinoma
* Computed tomography (CT) or magnetic resonance imaging (MRI) confirmed advanced ESCC which need neoadjuvant chemotherapy before surgical resection.
* Measurable disease according to the Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 criteria(diameter of the lesion should be more than 10mm by spiral CT or MRI, more than 20mm by common CT, the date of image should be less than 21 days before enrollment)
* Life expectancy of ≥3 month
* Eastern Cooperative Oncology Group (ECOG) 0-1
* Body Mass Index (BMI) ≥18.5kg/m2
* WBC>3,000/mm3, absolute neutrophil count ≥1500/mm3, platelet>100,000/mm3, Hb>9g/dl，Bilirubin level < 1.5 times ULN，Serum creatinine <1.5 times ULN，ALT and AST<2.5 times ULN ，AKP < 2.5 times ULN ，(≤5 times ULN in patients with liver metastases)(within 7 days before enrollment)
* No sever complication, such as active gastrointestinal bleeding, perforation, jaundice, obstruction, non-cancerous fever>38℃.
* Good compliance

Exclusion Criteria:

* Have used metformin or biguanide in the past
* Contraindications of metformin
* Unable to take metformin orally because of esophageal stenosis
* Currently receiving other effective regimens
* Previous anticipate other clinical trial within 4 weeks before entering this study
* No measurable lesions, eg. pleural fluid and ascites\
* Only with other previous malignancy within 5 year, except non-melanoma skin cancer and cervical carcinoma in situ
* Heart failure or other sever organ dysfunction, eg. coronary artery disease, myocardial infarction within the last 6 months only Brain or bone metastasis
* Mentally abnormal or disable cognition,including central nervous system (CNS) metastasis
* HIV infection, active hepatitis B or hepatitis C
* Unstable systemic diseases such as poorly controlled diabetes
* Interstitial lung disease, such as interstitial pneumonia, pulmonary fibrosis, or evidence of interstitial lung disease showed in X-ray/CT
* Known hypersensitivity to study drugs
* Pregnancy or lactation period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-02-05 (Estimated); Primary Completion 2020-03-20 (Estimated); Study Completion 2020-06-20 (Estimated)

PRIMARY OUTCOMES:
Tumor metabolic pathway | Through study completion, an average of 1 year
  To compare the changes of tumor metabolic pathway of pre-chemotherapy endoscopic biopsy samples and post-chemotherapy surgical resection samples
Tumor microenvironment | Through study completion, an average of 1 year
  To compare the changes of tumor microenvironment of pre-chemotherapy endoscopic biopsy samples and post-chemotherapy surgical resection samples

SECONDARY OUTCOMES:
Rate of pathologic complete response（pCR） | Through study completion, an average of 1 year
  Rate of pathologic complete response

CONTACTS AND LOCATIONS:
Overall Officials: Zhihao Lu, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Peking Universtiy Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No